CLINICAL TRIAL: NCT00961701
Title: Atherogenic Lipoprotein Phenotype and LDL Size and Subclasses in Patients With Primary Hyperparathyroidism
Brief Title: Lipids Profile in Primary Hyperparathyroidism
Acronym: LPHP
Status: Terminated | Type: Observational
Why Stopped: sample size was not enrolled
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: University of Palermo (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, avraham ishay, Dr, HaEmek Medical Center, Israel
Other Study IDs: 0097.09EMC
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe Primary hyperparathyroidism (PHP) has been associated with increased cardiovascular morbidity and mortality. Hypertension, dyslipidemia and impaired glucose tolerance were demonstrated in severe PHP, with improvement after surgery in these variables. Recent evidence suggests that the 'quality' rather than only the 'quantity' of low-density lipoprotein (LDL)-cholesterol exerts a direct influence on the cardiovascular risk. Thus, the proposed study protocol is intended to evaluate lipoprotein phenotype and LDL size and subclasses in patients with primary hyperparathyroidism.

DETAILED DESCRIPTION:
Severe traditional PHP has been associated with increased cardiovascular morbidity and mortality with an increase in acute MI prior to surgery.PHP is associated with increased prevalence of left ventricular hypertrophy, independent of blood pressure. Also prevalent in PHP, are valvular and myocardial calcifications as well as diastolic filling impairment, with a significant correlation with serum calcium and PTH levels.

Hypertension, dyslipidemia and impaired glucose metabolism were demonstrated in severe PHP, with improvement after surgery in these variables.Glucose tolerance test performed in patients with PHP revealed that 51% had impaired glucose tolerance, 34% had diabetes mellitus and 17% had impaired fasting glucose values. After successful parathyroidectomy fasting and 2-h plasma glucose falls significantly. Others have demonstrated hyperinsulinemia and impaired glucose tolerance without normalization after parathyroidectomy.

Most of the literature showing an increased cardiovascular risk is in those patients with more severe PHP .Patients with mild PHP had higher serum cholesterol, triglycerides, glucose, urate and hemoglobin values compared with controls.Also, moderate to severe vitamin D deficiency is a risk factor for developing cardiovascular disease especially in patients with hypertension.

Atherosclerosis is a diffuse disease formerly considered a lipid storage disease, which actually involves an ongoing inflammatory response. Elevated circulating levels of acute phase proteins, cytokines, and cell adhesion molecules indicate that inflammatory processes are occurring systemically . C-reactive protein [CRP] and the presence of metabolic syndrome were interrelated and were highly predictive for cardiovascular disease. Hyperinsulinemia was proposed as the common factor of all the traditional risk factors for cardiovascular disease, and insulin resistance is recognized as a chronic low-level inflammatory state.Although various inflammatory markers were individually significantly related to future cardiovascular disease risk, they added very little additional prognostic information to the traditional markers.

Recently, we have shown that greater probability of metabolic syndrome and insulin resistance were observed in patients with severe PHP. Serum calcium is a predictor of these cardiovascular risk factors.

Recent evidence suggests that the 'quality' rather than only the 'quantity' of LDL exerts a direct influence on the cardiovascular risk. LDL comprises multiple distinct subclasses that differ in size, density, physicochemical composition, metabolic behaviour and atherogenicity. There are at least four major subspecies of LDL (e.g. large LDL-I, medium LDL-II, small LDL-III, very small LDL-IV) and the predominance of small dense LDL has been accepted as an emerging cardiovascular risk factor .

Thus, the proposed study protocol is intended to evaluate lipoprotein phenotype and LDL size and subclasses in patients with primary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hyperparathyroidism

Exclusion Criteria:

* pregnant women
* patient taking hypolipidemic drugs
* patients with known cardiovascular, peripheral or cerebral atherosclerotic disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at the Endocrine Institute
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2016-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Luboshitzky, MD, Study Director — Endocrine Institute, Haemek Medical Center, Afula, Israel; Manfredi Rizzo, MD, Study Chair — University of Palermo; Giatgen Spinas, MD, Study Chair — University of Zurich; Kaspar Berneis, MD, Study Chair — University of Zurich
Locations (1):
- Endocrine Institute , Haemek Medical Center, Afula, Israel